CLINICAL TRIAL: NCT03055286
Title: A Phase 1b/2a Clinical Study of CWP232291 in Combination With Cytarabine in Subjects With Relapsed or Refractory Acute Myeloid Leukemia (AML)
Brief Title: Clinical Study of CWP232291 in Acute Myeloid Leukemia Patients
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: business/strategic reason
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JW-231A-103
Record Dates: First submitted 2017-02-03; First posted 2017-02-16 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CWP232291 in combination with cytarabine (ara-C) (Experimental)
  Interventions: Drug: CWP232291

INTERVENTIONS:
Drug: CWP232291 — For cohort 1-3, a fixed dose of ara-C at 1 G/m2 will be administered IV over 2 hours daily from Day 1 to Day 5 following CWP232291 infusion.
  For cohort 4, a fixed dose of ara-C at 1 G/m2 will be administered IV over 2 hours daily from Day 1 to Day 7 following 250 mg/m2 CWP232291 infusion.

SUMMARY:
This is a multicenter (S. Korea/US), Phase Ib, open-label, dose-finding study to assess safety, PK, PD, and preliminary efficacy of CWP232291 administered in combination with ara-C in subjects with relapsed or refractory AML.

The primary objectives in phase 2a is to assess the efficacy of CWP232291 administered in combination with cytarabine (response rate complete remission [RR-CR]/complete remission with incomplete blood count recovery [CRi]/partial remission [PR]).

ELIGIBILITY:
Inclusion Criteria:

1. Understands and is willing to sign an informed consent form (ICF) prior to initiation of any study-specific procedure.
2. 18 years of age at the time of consenting.
3. A pathologically confirmed diagnosis of AML by World Health Organization (WHO) classification that is progressing.
4. Has failed (refractory) or relapsed after no more than 2 prior regimens, and for whom for whom no other standard therapy options are available.
5. Subjects with prior autologous and allogeneic hematopoietic stem cell transplantation (allo HSCT) are eligible.
6. Adequate laboratory results including the following:

   * Serum creatinine ≤ 2.0 mg/dL
   * Total bilirubin ≤ 1.5 x upper limit of institutional normal (ULN), unless due to Gilbert's syndrome
   * Aspartate transaminase (AST) or alanine transaminase (ALT) ≤ 3 x ULN, unless due to organ leukemic involvement
7. Eastern Cooperative Oncology Group (ECOG) performance score 0-2.
8. The subject should be off any anticancer therapy including chemotherapy, immunotherapy, radiotherapy, hormonal, biologic or any investigational agents for at least 14 days or 5 half lives, whichever is greater, prior to enrollment with the exception of hydroxyurea. All prior treatment-related non-hematologic toxicities must have resolved to ≤ grade 2 prior to screening.
9. Female subject of childbearing potential (ie, premenopausal or not surgically sterile) must agree to use effective contraception from Day 1 until 28 days after the last dose of study drug, and have a negative serum or urine pregnancy test within 2 weeks prior to Day 1. Sexually active male subjects must also use effective contraception from Day 1 until 90 days after the last dose of any study drug.
10. Female subject must agree not to breastfeed at screening and throughout the study period and for 45 days after the final study drug administration. Female subject must not donate ova starting at screening and throughout the study period and for 45 days after the final study drug administration.
11. Male subject must not donate sperm starting at screening and throughout the study period and for 90 days after the final study drug administration.
12. Agree to adhere to all study protocol requirements.

Exclusion Criteria:

1. Subject has BCR-ABL-positive leukemia (Chronic myeloid leukemia [CML] in blast crisis).
2. Subject is diagnosed as acute promyelocytic leukemia (APL).
3. Subject has AML secondary to prior chemotherapy.
4. Subject has active clinically significant graft versus host disease (GVHD) or is on treatment with systemic corticosteroids for GVHD (except grade 1 skin GVHD). At least 3 months must have elapsed since completion of allogeneic stem cell transplantation.
5. Subject had a myocardial infarction within 6 months of enrollment, heart failure (New York Heart Association (NYHA) Class III or IV), uncontrolled angina, severe uncontrolled ventricular arrhythmias, left ventricular ejection fraction (LVEF) ≤ 40% or evidence of acute ischemia or active conduction system abnormalities.
6. Presence of a systemic fungal, bacterial, viral or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment).
7. Known in tolerance and allergy to cytarabine.
8. Active central nervous system (CNS) disease.
9. Known positive status for human immunodeficiency virus (HIV) and/or active hepatitis B or C.
10. Prior exposure to CWP232291.
11. Pregnant or breastfeeding women.
12. Suitable for imminent bone marrow transplant, or within 4 weeks of one.
13. Major surgery within 4 weeks prior to the first study dose.
14. Concurrent other malignancy, unless the patient has been disease-free for at least five years following curative intent therapy, with the following exceptions: (1) adequately treated in-situ carcinoma of cervix; (2) localized basal cell or squamous cell carcinoma of skin; (3) previous malignancy confined and treated locally (surgery or other modality) with curative intent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2025-08-26 (Actual); Study Completion 2025-08-26 (Actual)

PRIMARY OUTCOMES:
Recommended Phase 2 dose | up to 4 weeks
  To be determinded Recommended Phase 2 dose (RP2D) of CWP232291 in combination with cytarabine (ara-C), administered to subjects with relapsed or refractory AML.

SECONDARY OUTCOMES:
Cmax as a Pharmacokinetic (PK) assessments for CWP232291 | 3rd Cycle (each cycle = 28 days), Cycle 1 Day 1: Pre, 0.5hr, 1hr, 2hr, 3hr, 4hr, 5hr, 8hr, and 24hr after the start of infusion in Part A and at Cycle 1 Day 1: Pre, 2hr, 4hr, 8hr, and 24hr after the start of infusion in Part B.
  maximum plasma concentration (Cmax)
tmax as a Pharmacokinetic (PK) assessments for CWP232291 | 3rd Cycle (each cycle = 28 days), Cycle 1 Day 1: Pre, 0.5hr, 1hr, 2hr, 3hr, 4hr, 5hr, 8hr, and 24hr after the start of infusion in Part A and at Cycle 1 Day 1: Pre, 2hr, 4hr, 8hr, and 24hr after the start of infusion in Part B.
  time to maximum observed plasma concentration (tmax)
AUC0-t as a Pharmacokinetic (PK) assessments for CWP232291 | 3rd Cycle (each cycle = 28 days), Cycle 1 Day 1: Pre, 0.5hr, 1hr, 2hr, 3hr, 4hr, 5hr, 8hr, and 24hr after the start of infusion in Part A and at Cycle 1 Day 1: Pre, 2hr, 4hr, 8hr, and 24hr after the start of infusion in Part B.
  area under the time-concentration curve from time zero to the last measurable concentration (AUC0-t)
AUC0-∞ as a Pharmacokinetic (PK) assessments for CWP232291 | 3rd Cycle (each cycle = 28 days), Cycle 1 Day 1: Pre, 0.5hr, 1hr, 2hr, 3hr, 4hr, 5hr, 8hr, and 24hr after the start of infusion in Part A and at Cycle 1 Day 1: Pre, 2hr, 4hr, 8hr, and 24hr after the start of infusion in Part B.
  area under the time concentration curve from time zero to infinity (AUC0-∞)
AUC0-τ as a Pharmacokinetic (PK) assessments for CWP232291 | 3rd Cycle (each cycle = 28 days), Cycle 1 Day 1: Pre, 0.5hr, 1hr, 2hr, 3hr, 4hr, 5hr, 8hr, and 24hr after the start of infusion in Part A and at Cycle 1 Day 1: Pre, 2hr, 4hr, 8hr, and 24hr after the start of infusion in Part B.
  area under the time concentration curve from time zero the end of the dosage interval (AUC0-τ)
t½ as a Pharmacokinetic (PK) assessments for CWP232291 | 3rd Cycle (each cycle = 28 days), Cycle 1 Day 1: Pre, 0.5hr, 1hr, 2hr, 3hr, 4hr, 5hr, 8hr, and 24hr after the start of infusion in Part A and at Cycle 1 Day 1: Pre, 2hr, 4hr, 8hr, and 24hr after the start of infusion in Part B.
  terminal elimination half-life (t½)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (2):
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Washington, Seattle, Washington
- South Korea (3):
  - Samsung medical center, Seoul, Gangnam-gu
  - Seoul National University Hospital, Seoul, Jongno-gu
  - Asan Medical Center, Seoul, Songpa-Gu